CLINICAL TRIAL: NCT02741622
Title: Effects of Aerobic Exercise Intensity on Affective States and Brain Derived Neurotropic Factor in Patients With Depression
Brief Title: Brain Derived Neurotropic Factor Response to Aerobic Exercise Intensity in Depressive Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/2230
Record Dates: First submitted 2016-03-15; First posted 2016-04-18 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Depressive Disorder; Depressive Disorder, Major
Keywords: Exercise therapy
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Acute High aerobic intensity training (HIT) and long slow distance training (LSD)
  Interventions: Behavioral: High aerobic intensity training (HIT); Behavioral: Long slow distance training (LSD)

INTERVENTIONS:
Behavioral: High aerobic intensity training (HIT) — One training session, high aerobic intensity training (HIT) at 90-95 % of the maximal heart rate (HRmax)
Behavioral: Long slow distance training (LSD) — One training session, long slow distance training (LSD) at 70 % of the HRmax

SUMMARY:
Acute aerobic exercise improves affective stats in patients with mental illnesses. Brain derived neurotropic factor (BDNF) may be a biological mechanism that contributes to the affective benefits. The magnitude of the increase of serum BDNF might be exercise intensity dependent, but no study has compared low high-aerobic-intensity training at 90-95 % of the maximal heart rate (HRmax) with long-slow-distance training at 70 % of the HRmax in patients with depression.

The aim of this study is to compare changes in serum BDNF levels after high-aerobic-intensity training and long-slow-distance training in a intra-individual design in patients suffering from depression. The results will give indications of a possible difference in BDNF response between aerobic intensities and may be uses as pilot data for calculating sample size.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe depression (ICD10: F32-F33)

Exclusion Criteria:

* Bipolar disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in serum brain derived neurotropic factor (BDNF) | 15 minutes before exercise to 5> minutes after exercise.
  To measure serum BDNF levels, blood samples will be taken before and after each workout session.

SECONDARY OUTCOMES:
Change in affective symptoms | 15 minutes before exercise to 15> minutes after exercise.
  The positive and negative affect schedule (PANAS) .
Change in state of anxiety. | 15 minutes before exercise and 15> minutes after exercise.
  A short form of state trait anxiety inventory for adults (STAI) is used to detect their state of anxiety.
Change in subjective exercise experience | 15 minutes before exercise to 15> minutes after exercise.
  The Subjective exercise experience scale (SEES).
Maximal oxygen uptake | Baseline
Maximal Heart rate | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pål Sandvik, MD, Study Director — St.Olavs University Hospital, Østmarka
Locations (1):
- St.Olavs university Hospital, Departement of Østmarka, Trondheim, Norway